CLINICAL TRIAL: NCT00619567
Title: Pilot Study of an Internet-Based Cognitive Stimulation Program in AIDS
Brief Title: Cognitive Stimulation Program in AIDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SB1723; R03MH081723-01 (NIH)
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: Cognition; Rehabilitation; Cognitive Stimulation; Human Immunodeficiency Virus; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Stimulation (Experimental): Subjects will be given Internet access to the Smartbrain cognitive stimulation program. They will complete exercises for ~30 minutes, at least three times per week, for a period of 24 weeks.
  Interventions: Behavioral: Smartbrain
- Control (No Intervention): These individuals will receive "usual care" during the 24 week follow-up period.

INTERVENTIONS:
Behavioral: Smartbrain — The initial session will be set for 10 minutes, with weekly increases (of 10 minutes) to a maximum of 30 minutes per day, 7 days a week. Each subject will be trained using the same modules of the Smartbrain protocol, with an emphasis on speed of information processing.
  Other Names: Cognitive stimulation
  Arms: Cognitive Stimulation

SUMMARY:
There has been little success in treating the cognitive (thinking) problems associated with HIV/AIDS using medications. The purpose of this study is to determine whether an internet-based cognitive "stimulation" program might help HIV-infected individuals think more clearly. If this is true, then it means that people with mild forms of cognitive impairment may be able to help themselves to get better.

DETAILED DESCRIPTION:
The neurocognitive manifestations of HIV/AIDS have long been recognized as important for the management, survival, and quality of life of affected patients and their families. Following the advent of Highly active anti-retroviral therapy (HAART) the incidence of HIV-associated dementia (HAD) has fallen, but the prevalence of the milder forms of HIV-related cognitive disorders has risen. This is important because alterations in cognitive function can have significant impact on work and social activities, mood, and perceived quality of life. To date, pharmacological management of HIV-associated cognitive disorders - apart from HAART - have met with limited success (e.g., Peptide T, Ritalin). Therefore, it appears reasonable to ask whether the use of non-pharmacological tools might help alleviate or ameliorate the symptoms of the milder forms of cognitive impairment, and thus improve mood and activities of daily living. The purpose of this application is to request funds to allow us to complete a feasibility/pilot study of the merits of using an internet-based cognitive stimulation program (CSP) to improve the cognitive functions and quality of life of individuals with HIV/AIDS, and, secondarily, to detect such changes using a computerized assessment tool designed for use in a health care practitioner's office (Computer-Based Assessment of Mild Cognitive Impairment (CAMCI)).

ELIGIBILITY:
Inclusion Criteria:

* Access to the Internet (either from home or public access)
* Native language is English
* HIV infected

Exclusion Crieria:

* Active drug/alcohol abuse or dependence
* Current major depression
* History of neurological disease, Central Nervous System Opportunistic Infections, tumors, or stroke
* History of learning disability or Attention Deficit/Hyperactivity Disorder (by subject report).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Global Impairment Rating from battery of neuropsychological tests. | 24 weeks

SECONDARY OUTCOMES:
Change in perceived quality of life using MOS/HIV | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James T. Becker, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, University of Pittsburgh, Pittsburgh, Pennsylvania, United States